CLINICAL TRIAL: NCT02432612
Title: An Open-label, Multi-centre, Single-dose Clinical Trial to Assess the Pharmacokinetic (PK) Properties and Tolerability of a Single Oromucosal Dose of 6 Sprays of Sativex® in Patients With Advanced Cancer Currently on Background Step III Opioid Therapy
Brief Title: A Study to Assess the Pharmacokinetic (PK) Properties of Sativex® in Patients With Advanced Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Organization: GWPharm (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWCP1450
Record Dates: First submitted 2015-03-26; First posted 2015-05-04 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sativex (Experimental): Sativex will be administered by trained, clinical trial personnel, via a pump action oromucosal spray. Sativex will be administered as 2 actuations (sprays) under the tongue or inside the cheeks every 4 minutes until 6 sprays have been administered. Following the administration of the first and second set of 2 actuations, patients will be offered 50 mL water to drink; and following the final set of 2 actuations, 100 mL of water will be offered (i.e., a total of 200 mL water will be offered during the Sativex dosing). There must be a period of at least 2 minutes and no more than 3 minutes between Sativex administration and consumption of water. Patients will not be permitted their regular medication until 2 hours post dose of investigational medicinal product (IMP) to minimize any possible drug interactions.
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: Sativex — Sativex is supplied as a liquid containing 27 mg/mL Δ9-tetrahydrocannabinol (THC) and 25 mg/mL Cannabidiol (CBD) plus peppermint flavoring. Each 100 µL actuation of the pump-action spray delivers 100 µL 27 mg THC and 25 mg CBD.
  Other Names: Nabiximols; GW-1000-02; THC/CBD spray

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of a single oromucosal dose of Sativex in subjects with advanced cancer currently on background Step III opioid therapy.

DETAILED DESCRIPTION:
This is an open-label, multiple-centre, single dose clinical trial to assess the PK of a single oromucosal dose of Sativex in subjects with advanced cancer who are currently on background Step III opioid therapy.

A minimum of 25 subjects ≥18 years with advanced cancer will be needed for the assessment of the primary objective of the trial. The Screening Visit (Visit 1) will be performed within -10 to -2 days prior to dosing. For the Screening Visit, subjects will attend on an outpatient basis.

Subjects will be checked into the clinical research facility on Day -1 and will be confined to the clinical research facility for the Inpatient/Treatment Period (Day -1 to Day 3) (Visit 2). Subjects will be administered a single oromucosal dose of Sativex on Day 1 (time [t]=0). Fourteen PK blood samples will be taken from Day 1 to Day 3 during Visit 2: one predose sample and 13 postdose samples at the following time points after dosing: 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours postdose.

Subjects will be discharged from the clinical research facility after the 48-hour PK blood sample has been taken and final safety assessments are completed. Subjects who discontinue from the trial prior to the completion of the PK blood draws will undergo the safety evaluations scheduled for Day 3.

The Safety Follow-up Call (Visit 3) will be made 7 (+2) days after dosing on Day 1. Subjects with any new adverse events (AEs) or clinical laboratory abnormalities will be asked to return for safety follow-up.

The expected duration for trial participation (including Screening Visit, Inpatient/Treatment Period, and Safety Follow-up Call) for each individual subject is a maximum of 19 days.

ELIGIBILITY:
For inclusion in the trial subjects must fulfil ALL of the following criteria:

* The subject is aged ≥18 years.
* The subject has advanced cancer for which there is no known curative therapy.
* The subject has a clinical diagnosis of cancer related pain, is currently taking Step III opioid therapy and is willing to continue on their current dosing regimen throughout the Inpatient/Treatment Period of the trial.
* The subject is willing and able to give written informed consent.
* The subject is willing and able to comply with all trial requirements.

The subject may not enter the trial if ANY of the following apply:

* The subject is receiving intrathecal opioids via pump mechanism.
* The subject is currently using or has used cannabis or cannabinoid based medications within 30 days of trial entry and is unwilling to abstain for the duration of the trial.
* The subject has any known or suspected history of a substance abuse/dependence disorder (including opiate abuse/dependence prior to the diagnosis of cancer); current heavy alcohol consumption (more than 60 grams of pure alcohol per day for men, and more than 40 grams of pure alcohol per day for women) and unwilling to abstain from alcohol for 24 hours prior to and during trial visits; current use of an illicit drug or current non prescribed use of any prescription drug.
* The subject has a history of epilepsy as evidenced by one or more seizures in the last 12 months.
* The subject has any known or suspected history or family history of schizophrenia, or other psychotic illness, history of severe personality disorder or other severe significant psychiatric disorder other than depression associated with the underlying condition.
* The subject has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP.
* The subject has significant cardiac disease, or has a cardiac disorder that in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction, or has a secondary or tertiary atrioventricular block, or evidence of clinically significant cardiac disease on ECG at the Screening Visit.
* The subject has significantly impaired renal function as evidenced by a creatinine clearance (based on measured serum creatinine level) lower than 40 mL/min at Visit 1.
* The subject has significantly impaired hepatic function at Visit 1 (alanine aminotransferase [ALT] >5 upper limit of normal (ULN) or total bilirubin [TBL] > 2 ULN). If the ALT or aspartate aminotransferase [AST] >3 ULN and the TBL >2 ULN [or international normalized ratio [INR] >1.5]) this subject must not enter the trial.
* The subject is a female of childbearing potential, or a male patient whose partner is of childbearing potential, is unwilling to ensure that they and/or their partner use a highly effective method of contraception, including female sterilization (ie, documented bilateral tubal ligation), male sterilization, established use of hormonal methods of contraception (oral, implanted or transdermal), an intrauterine device or intrauterine system, or true abstinence.
* Female subject who is pregnant, lactating or planning pregnancy during the course of the trial and for 3 months thereafter.
* The subject has received a non approved IMP within 30 days or 5 times the half-life of the IMP (whichever is greater) prior to the Screening Visit.
* The subject has any other significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the trial, or may influence the result of the trial, or the patient's ability to participate in the trial.
* The subject was previously enrolled in the current trial or any other Sativex clinical trial for cancer pain.
* The subject is unwilling to abstain from the consumption of grapefruit products during the week prior to and throughout the Inpatient/Treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic endpoints of the analyte delta 9-tetrahydrocannabinol (THC). | 0-48 hours post-dose
  • Mean maximum plasma concentration (Cmax) of THC.
Pharmacokinetic endpoints of the analyte THC. | 0-48 hours post-dose
  • Mean area under the concentration-time curve calculated from time zero to the last observable concentration at time t (AUC(0-t)) of THC.
Pharmacokinetic endpoints of the analyte THC. | 0-48 hours post-dose
  • Mean area under the concentration-time curve from time zero to infinity (AUC(0-∞)) of THC.
Pharmacokinetic endpoints of the analyte 11-hydroxy-delta 9-tetrahydrocannabinol (11-OH-THC). | 0-48 hours post-dose
  • Mean Cmax of 11-OH-THC.
Pharmacokinetic endpoints of the analyte 11-OH-THC. | 0-48 hours post-dose
  • Mean AUC(0-t)) of 11-OH-THC.
Pharmacokinetic endpoints of the analyte 11-OH-THC. | 0-48 hours post-dose
  • Mean AUC(0-∞) of 11-OH-THC.
Pharmacokinetic endpoints of the analyte 11-carboxy-delta 9-tetrahydrocannabinol (11-COOH-THC). | 0-48 hours post-dose
  • Mean Cmax of 11-COOH-THC.
Pharmacokinetic endpoints of the analyte 11-COOH-THC. | 0-48 hours post-dose
  • Mean AUC(0-t)) of 11-COOH-THC.
Pharmacokinetic endpoints of the analyte 11-COOH-THC. | 0-48 hours post dose
  • Mean AUC(0-∞) of 11-COOH-THC.
Pharmacokinetic endpoints of the analyte cannabidiol (CBD). | 0-48 hours
  • Mean Cmax of CBD.
Pharmacokinetic endpoints of the analyte CBD. | 0-48 hours
  • Mean AUC(0-t) of CBD.
Pharmacokinetic endpoints of the analyte CBD. | 0-48 hours
  • Mean AUC(0-∞) of CBD.
Pharmacokinetic endpoints of the analyte 6-hydroxy-cannabidiol (6-OH-CBD). | 0-48 hours.
  • Mean Cmax of 6-OH-CBD.
Pharmacokinetic endpoints of the analyte 6-OH-CBD. | 0-48 hours
  • Mean AUC(0-t) of 6-OH-CBD.
Pharmacokinetic endpoints of the analyte 6-OH-CBD. | 0-48 hours.
  • Mean AUC(0-∞) of 6-OH-CBD.
Pharmacokinetic endpoints of the analyte 7-hydroxy-cannabidiol (7-OH-CBD). | 0-48 hours
  • Mean Cmax of 7-OH-CBD.
Pharmacokinetic endpoints of the analyte 7-OH-CBD. | 0-48 hours
  • Mean AUC(0-t) of 7-OH-CBD.
Pharmacokinetic endpoints of the analyte 7-OH-CBD. | 0-48 hours
  • Mean AUC(0-∞) of 7-OH-CBD.
Pharmacokinetic endpoints of the analyte 7-carboxy-cannabidiol (7-COOH-CBD). | 0-48 hours
  • Mean Cmax of 7-COOH-CBD.
Pharmacokinetic endpoints of the analyte 7-COOH-CBD. | 0-48 hours
  • Mean AUC(0-t) of 7-COOH-CBD.
Pharmacokinetic endpoints of the analyte 7-COOH-CBD. | 0-48 hours
  • Mean AUC(0-∞) of 7-COOH-CBD.

SECONDARY OUTCOMES:
Pharmacokinetic endpoints of the analyte THC. | 0-48 hours post-dose
  • Mean half-life (t1/2) of THC.
Pharmacokinetic endpoints of the analyte THC. | 0-48 hours post-dose
  • Mean time to maximum plasma concentration (tmax) of THC.
Pharmacokinetic endpoints of the analyte THC. | 0-48 hours post-dose
  • Mean apparent clearance of drug from plasma after extravascular administration (CL/F) of THC.
Pharmacokinetic endpoints of the analyte THC. | 0-48 hours post-dose
  • Mean apparent volume of distribution (Vd/F) of THC.
Pharmacokinetic endpoints of the analyte 11-OH-THC. | 0-48 hours post-dose
  • Mean t1/2 of 11-OH-THC.
Pharmacokinetic endpoints of the analyte 11-OH-THC. | 0-48 hours post-dose
  • Mean tmax of 11-OH-THC.
Pharmacokinetic endpoints of the analyte 11-COOH-THC. | 0-48 hours post-dose
  • Mean t1/2 of 11-COOH-THC.
Pharmacokinetic endpoints of the analyte 11-COOH-THC. | 0-48 hours post-dose
  • Mean tmax of 11-COOH-THC.
Pharmacokinetic endpoints of the analyte CBD. | 0-48 hours post-dose
  • Mean t1/2 of CBD.
Pharmacokinetic endpoints of the analyte CBD. | 0-48 hours post-dose
  • Mean tmax of CBD.
Pharmacokinetic endpoints of the analyte CBD. | 0-48 hours post-dose
  • Mean CL/F of CBD.
Pharmacokinetic endpoints of the analyte CBD. | 0-48 hours post-dose
  • Mean Vd/F of CBD.
Pharmacokinetic endpoints of the analyte 6-OH-CBD. | 0-48 hours post-dose
  • Mean t1/2 of 6-OH-CBD.
Pharmacokinetic endpoints of the analyte 6-OH-CBD. | 0-48 hours post-dose
  • Mean tmax of 6-OH-CBD.
Pharmacokinetic endpoints of the analyte 7-OH-CBD. | 0-48 hours post-dose
  • Mean t1/2 of 7-OH-CBD.
Pharmacokinetic endpoints of the analyte 7-OH-CBD. | 0-48 hours post-dose
  • Mean tmax of 7-OH-CBD.
Pharmacokinetic endpoints of the analyte 7-COOH-CBD. | 0-48 hours post-dose
  • Mean t1/2 of 7-COOH-CBD.
Pharmacokinetic endpoints of the analyte 7-COOH-CBD. | 0-48 hours post-dose
  • Mean tmax of 7-COOH-CBD.
The incidence of adverse events as a measure of subject safety. | From screening to follow-up (a maximum of 19 days).
  The number of subjects who experienced an adverse event during the study is presented. The time-frame for adverse event reporting was from screening to follow-up visit.
The number of subjects with a clinically significant change in physical and oral examination results, relative to pre-treatment baseline. | From screening to follow-up (a maximum of 19 days)
  The number of subjects with a change in physical and oral examination results indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with a clinically significant change in in 12-lead ECG (electrocardiogram) results, relative to pre-treatment baseline. | From screening to follow-up (a maximum of 19 days)
  The number of subjects with a change in ECG results indicative of an adverse event, relative to the pre-treatment baseline, is presented.
The number of subjects with clinically significant changes in laboratory test parameters, relative to pre-treatment baseline. | From screening to follow-up (a maximum of 19 days)
  The number of subjects with clinically significant changes in serum biochemistry, haematology and urinalysis, relative to the pre-treatment baseline, is presented.
The number of subjects with a clinically significant change in vital signs, relative to pre-treatment baseline. | From screening to follow-up (a maximum of 19 days)
  The number of subjects with a clinically significant change in vital signs (supine/sitting blood pressure and pulse rate) indicative of an adverse event relative to the pre-treatment baseline, is presented.